CLINICAL TRIAL: NCT07235332
Title: Assessment of Exposure to Toxic Metals in Relation to Different Diet Patterns - the DietBiom CALC-M Study: Dietary Biomonitoring of Cadmium, Arsenic, Lead, Chromium, and Mercury
Brief Title: Assessing Toxic Metal Exposure From Vegetarian/Vegan, Omnivorous, and Low-carb Diets in Israel.
Status: Enrolling by invitation | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: AU-HEA-AB-20240729
Record Dates: First submitted 2025-09-11; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Environmental Exposure; Dietary Patterns; Nutritional Epidemiology; Human Biomonitoring
MeSH Terms: interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — morning spot urine, serum and whole blood samples will be retained for optional future studies

GROUPS / COHORTS (3):
- omnivorous: Healthy adults aged 20-49 years who consume a regular mixed diet including both plant and animal foods. Participants must have maintained this diet pattern for ≥ 1 year prior to enrollment. Exclusion criteria include class 3 obesity (BMI ≥ 09.9 kg/m²), or any chronic illness. Participants will complete dietary questionnaires and provide biological samples for assessment of toxic-metal exposure and nutritional biomarkers.
  Interventions: Behavioral: Screening
- low carb: Healthy adults aged 20-49 years adhering for ≥ 1 year to a carbohydrate-restricted or animal-based diet, such as ketogenic, paleo, or carnivore-style patterns. Diets emphasize animal-derived foods and limit carbohydrate intake. Eligible participants have BMI 18.5-39.9 kg/m² and no chronic medical conditions. Group will undergo identical dietary, anthropometric, and biological assessments to quantify toxic-metal exposure and nutritional-status indicators.
  Interventions: Behavioral: Screening
- Plant based: Healthy adults aged 20-49 years who have followed a vegetarian or vegan diet for ≥ 1 year. Participants consume no meat, poultry, or fish; vegans avoid all animal products. The target composition is about 20 % vegans within the plant-based group. BMI 18.5-39.9 kg/m², and free of chronic disease. Participants will provide dietary data (FFQ + 3-day food record), anthropometric measurements, and biological samples for toxic-metal and nutritional-status assessment.
  Interventions: Behavioral: Screening

INTERVENTIONS:
Behavioral: Screening — no intervention. Just data collection in a cross-sectional study manner. We will collect blood and urine and preform BIA and DXA and also make them fill questioners

SUMMARY:
Different dietary intake may pose various health risks as as these have different potential exposure to heavy metals, which may originate from soils, irrigation systems, infrastructure, packaging, and other environmental exposures to toxic metals such as livestock nutritional intake. In this study, we aim to quantify toxic metals such as cadmium, lead, chromium, arsenic, and mercury, as well as macro and micronutrient contents in humans that are under three different diets (vegetarian-vegan, omnivorous, and low-carbohydrate diets). Short- and long-term nutritional intake will be obtained using food diaries and validated food frequency questionnaire, respectively. Analysis of essential nutrients as well as toxic metals will be assessed from nutritional software and database. Samples of blood (whole blood and serum) and urine as well as sub-samples of several common food items from 250 healthy volunteers will be collected and analyzed using standardized chemical protocol and quantified by an ICP-MS. Through the chemical results we intend to correlate dietary patterns with heavy metal exposure and identify diet-related exposure risks. These correlations will help in informing professionals and the public and will improve public health recommendations. This initiative stands out in its focus on a comprehensive dietary assessment to understand the impact of different dietary choices on metal exposure levels, particularly in the Israeli context.

DETAILED DESCRIPTION:
Detailed Study Description Sampling, Eligibility Criteria, and Sample Size

Participant recruitment will be initiated through social media campaigns targeting students from Ariel University and nearby academic institutions. Eligible participants will be healthy adults aged 20-45 years who have adhered for at least one year to one of three self-identified dietary patterns:

Plant-based diet (vegetarian or vegan; target 20% vegans),

Omnivorous diet ("regular" mixed diet), or

Low-carbohydrate diet (animal-based dietary patterns such as paleo or ketogenic).

Dietary pattern will be verified using a validated Food Frequency Questionnaire (FFQ) developed by the Israeli Ministry of Health, Department of Nutrition (adapted from Berman et al., 2023).

Exclusion criteria include obesity (BMI ≥ 30 kg/m²), underweight (BMI ≤ 18.5 kg/m²), or any chronic disease, verified via self-report and confirmed by a physician's medical summary.

Following informed consent, participants will complete the FFQ through the NutRatio® dietary-analysis software to confirm diet pattern. A brief phone interview and an instructional video will orient participants to study procedures and eligibility requirements.

We aim to recruit 250 participants in total, evenly distributed across the three diet groups. Participants will be frequency-matched by age (± 5 years), BMI (± 3 kg/m²), and smoking status, given smoking's established association with metal exposure. Sample size is based on ANOVA (Cohen's f = 0.25, medium effect size).

Measurement Day Protocol

Eligible participants will be scheduled for a standardized assessment session (~2 hours) at the MetaboLab, Department of Nutritional Sciences, Ariel University.

Short-term dietary intake: Participants will complete a 3-day food record (two weekdays + one weekend day) using NutRatio software within two weeks before their visit. The tool integrates USDA (SR-28), Israeli Ministry of Health (2017), and updated food label databases (2024). Participants will photograph each meal before and after eating, upload photos to the research team, and record foods immediately after consumption. The team will review entries daily, ensuring completeness and logical accuracy; missing or unclear data will be clarified by phone the next day.

NutRatio will quantify energy, macronutrients (including fatty-acid and amino-acid profiles), dietary fiber, selected vitamins (e.g., folate, B-12), and minerals (e.g., calcium, iron, zinc). Dietary metal exposure will be estimated from the reported foods using both NutRatio and additional reference databases. These values will later be compared to international toxicological thresholds (e.g., U.S. CDC, German Environment Agency).

Food Sampling for Toxic Metal Assessment

Based on correlations between reported intake and measured blood or urine metal levels, food groups most associated with each metal will be identified. Representative items will then be sampled for laboratory analysis.

For example, if mercury levels correlate strongly with fish intake, approximately six fish species or brands most commonly consumed by high-exposure participants will be purchased and analyzed. The type and brand of food will be confirmed through participant follow-up when necessary.

Each food item will undergo chemical digestion and quantification of metals (cadmium, lead, chromium, arsenic, mercury). Measured concentrations will be compared with international datasets including EFSA, Codex Alimentarius, U.S. NCEH, and the Israeli Ministry of Health (Food Control Services, 2016).

Anthropometric and Demographic Measures

Participants will attend the study visit after an overnight fast (water only). Measurements will include:

Weight and height (standardized protocols),

Body composition using InBody 570 (Biospace, Korea), a validated bioelectrical impedance analyzer providing body-fat, muscle-mass, and water-compartment data (Miller et al., 2016; Sirirat et al., 2020).

Questionnaires will collect demographic information, health history, smoking, occupational exposures (including military service), and lifestyle factors related to environmental pollutant exposure. These tools are adapted from Israel's national heavy-metal survey (Berman et al., 2023) and the European PARC initiative (https://www.eu-parc.eu

).

Biological Sample Collection and Chemical Analysis

Blood (whole and serum) and urine samples will be collected using BPA-free tubes and stored at -20 °C until analysis to prevent chemical degradation. Serum will be separated by controlled thawing (2-8 °C overnight), gentle mixing, clotting (30 min), centrifugation (15 min, 2000 rpm), and pipette aspiration. Whole-blood samples will be homogenized by vortex.

Samples (blood, serum, urine, and food) will be digested using analytical-grade nitric acid and hydrogen peroxide in a microwave digestion system following EPA 3052 protocols (Bocca et al., 2003). Blank samples will accompany each batch to determine limits of detection and quantification. Quality control will include certified reference materials and inter-laboratory validation using split samples.

Primary analyses will be conducted at Ariel University's Trace Metal Laboratory (Co-PI: Dr. Daniel Palchan). Additional or confirmatory analyses may occur at the Ministry of Health laboratory (Dr. Tamar Berman), Hebrew University, Weizmann Institute, or Geological Survey of Israel, depending on instrument availability.

Trace-element quantification will be performed using Inductively Coupled Plasma-Mass Spectrometry (ICP-MS) according to validated methods (Laur et al., 2020). Analytical protocols will align with CDC DLS 3040.1-01. Metal concentrations in blood and urine will be compared with reference values from national (Berman et al., 2023) and international surveys (CDC 2018; EFSA 2010; German Environment Agency 2023).

Results will be evaluated against Human Biomonitoring (HBM-I, HBM-II) thresholds (German Environment Agency 2023). Creatinine will be measured for urinary normalization.

Data Integration and Statistical Analysis

All data sources-FFQ, 3-day food record, anthropometric measures, biological samples, and chemical analyses-will be integrated into a unified database. Statistical analyses will examine relationships between dietary pattern and biomarker concentrations using ANOVA, multivariable regression, and correlation analyses. Dietary estimates of metal exposure will be compared with both measured biological levels and concentrations found in representative food samples.

Potential confounders (age, BMI, smoking, and occupational exposure) will be adjusted for in multivariate models. Sensitivity analyses will explore differences by sex and by vegan versus vegetarian subgroups within the plant-based group.

Pilot Study

A pilot phase involving 10 volunteers will precede full data collection. The pilot will test recruitment, informed-consent communication, FFQ completion, anthropometric assessment, biospecimen collection, and data-entry logistics. It will also be used to optimize sample-preparation protocols in the Trace Metal Laboratory.

If full analytical workflows cannot yet be implemented, mock data for metal levels will be generated to validate database structure and preliminary statistical pipelines. Biological samples from the pilot will be stored frozen for later analysis once full ICP-MS procedures are operational.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 to 49 years
* Generally healthy
* Following a specific diet (vegetarian/vegan, low-carbohydrate, or omnivorous) for at least one year
* Completion of all required screenings, including questionnaires, blood tests, morning urine sample, BIA, and DXA

Exclusion Criteria:

* Pregnancy
* Chronic illness or history of cancer
* High risk of heavy metal exposure (based on occupational data)
* Age outside 20 to 49 years
* Body mass index (BMI) greater than 40 kg/m²
* Incomplete data submission

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will initiate participant recruitment through social media outreach, targeting students from Ariel University as well as other academic institutes and areas located nearby Ariel University (the operating institution of the study). Eligible participants who will sign informed consent include young adults (20-45 years), identifying as vegetarians/vegans ("plantbased diet"; aim for 20% vegans), omnivores ("regular diet"), or low-carbohydrate diet followers ("animal-based diet" such as paleo, ketogenic diets, etc.) and following these diets for a minimum of one year (the statement on the personal diet pattern will be verified by using by a validated food frequency questionnaire [FFQ]) developed by the Israeli Ministry of Health, Department of Nutrition (adapted from (Berman et al., 2023).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
elevated toxic metal concentrations in blood, serum or urine | At time of enrolment (single measurement during the recruitment visit, within 2 month of consent)

CONTACTS AND LOCATIONS:
Locations (1):
- Ariel University, Ariel, Israel